CLINICAL TRIAL: NCT02063035
Title: Topical Application of Tranexamic Acid to Reduce Postoperative Blood Loss in Posterior Approach Spinal Surgery
Brief Title: Effectiveness Study of the Drug Tranexamic Acid to Reduce Post-surgery Blood Loss in Spinal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Kirkham Wood, Associate Professor at Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2012P000266; 2012P000266 (Other: Massachusetts General Hospital IRB approved)
Record Dates: First submitted 2013-12-19; First posted 2014-02-14 (Estimated); Results first posted 2017-06-08 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Lumbar Spinal Stenosis; Thoracic Spinal Stenosis
Keywords: lumbar spine surgery; thoracic spine surgery
MeSH Terms: conditions — Spinal Stenosis | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tranexamic acid (Experimental): Participants undergoing spinal surgery will receive a single, topical dose of tranexamic acid. The surgeon will irrigate the study medication in the wound prior to closure, and aspirate it after five minutes. Drains will be placed after the study drug has been aspirated.
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): Participants undergoing spinal surgery will receive a single, topical dose of matching placebo. The surgeon will irrigate the study medication in the wound prior to closure, and aspirate it after five minutes. Drains will be placed after the study drug has been aspirated.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid — A single topical application of 3 grams (g) of Tranexamic acid in 100 milliliter (mL) saline.
  Other Names: Cyklokapron®
  Arms: Tranexamic acid
Drug: Placebo — A single topical application of matching placebo, which is 100 mL of normal saline.
  Arms: Placebo

SUMMARY:
Hypothesis: Topical application of Tranexamic acid into the surgical wound during spine surgery will decrease the overall blood loss post-operatively. This reduction in blood loss will reduce the need for transfusion. In addition it will also significantly reduce the cost of the surgical procedure.

Specific Aim 1: The goal of this study is to quantitatively assess whether topical application of tranexamic acid placed into the surgical wound during lumbar spine surgery will decrease post-operative blood loss, thus lowering the need for blood transfusions. By reducing the number of transfusions participants can avoid the well-known complications associated with them. The investigators do not plan on measuring serum tranexamic acid levels.

Several meta-analyses and level I studies have shown that intravenous (IV) administration of tranexamic acid is effective in reducing postoperative blood loss and the need for transfusion.

DETAILED DESCRIPTION:
Tranexamic acid, an antifibrinolytic agent, has been studied at great length across a myriad of medical specialties to reduce blood lost during these surgeries. Topical tranexamic acid administration reduces postoperative blood loss and proved safe in multiple types of surgeries -e.g. cardiothoracic, oral and maxillofacial, eye, ear and throat.(References: Fawzy and others [et al], Wong et al, Zufferey et al, Wang et al, Ipema et al).

Intravenous tranexamic acid administration has been shown to reduce postoperative blood loss and transfusion need in patients undergoing spinal surgery (Reference: Elwatidy et al). Some advocates have suggested that topical (i.e. local) administration might be preferred over intravenous application. Topical administration of tranexamic acid has some potential advantages as it leads to lower systemic absorption, and offers less concern over the risk of thromboembolic complications (References: Wong et al, Raveendran et al).

While systemic (intravenous) use of tranexamic acid has been studied in spine surgery, there has been little studied to show its effectiveness at reducing blood loss when used topically.

This study proposes to determine if the topical application of tranexamic acid into the surgical wound of posterior multi-level lumbar spine surgery will decrease postoperative blood loss, thus decreasing the need for potential transfusions. Tranexamic acid has been well documented for its safety and efficacy, the investigators believe that this agent will become an important tool to reduce the blood loss in spinal surgeries. It offers a reduction in blood loss and, ultimately, a decrease in the transfusion rates which pose risks to the subject and significant cost.

ELIGIBILITY:
Inclusion Criteria:

* 18-85 years, both male and female
* Undergoing elective multi-level spinal surgery with a posterior approach to the thoracolumbar spine.
* Negative pregnancy test

Exclusion Criteria:

* Allergy to tranexamic acid
* Preoperative anemia (Hemoglobin <11 grams per deciliter [g/dL] )
* Coagulopathy (preoperative platelet count <150,000, International Normalized Ratio >1.4, or Partial Thromboplastin Time > 1.5 times normal)
* History of deep vein thrombosis, stroke, or pulmonary embolism
* Pregnant or breast feeding
* Liver function tests 2 times the upper limit of normal, and those with creatine greater than 1.6 milligrams per deciliter (mg/dL)
* Infection
* Revision procedure in which the only procedure is removing instrumentation
* Renal impairment
* Dural tear

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2015-04-22 (Actual); Study Completion 2015-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirkham B Wood, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Orthopedic Spine, Boston, Massachusetts, United States

REFERENCES:
- [Background] Fawzy H, Elmistekawy E, Bonneau D, Latter D, Errett L. Can local application of Tranexamic acid reduce post-coronary bypass surgery blood loss? A randomized controlled trial. J Cardiothorac Surg. 2009 Jun 18;4:25. doi: 10.1186/1749-8090-4-25. PMID 19538741
- [Background] Gill JB, Chin Y, Levin A, Feng D. The use of antifibrinolytic agents in spine surgery. A meta-analysis. J Bone Joint Surg Am. 2008 Nov;90(11):2399-407. doi: 10.2106/JBJS.G.01179. PMID 18978408
- [Background] Thompson GH, Florentino-Pineda I, Poe-Kochert C. The role of amicar in decreasing perioperative blood loss in idiopathic scoliosis. Spine (Phila Pa 1976). 2005 Sep 1;30(17 Suppl):S94-9. doi: 10.1097/01.brs.0000175188.05542.a9. PMID 16138073
- [Background] Hynes MC, Calder P, Rosenfeld P, Scott G. The use of tranexamic acid to reduce blood loss during total hip arthroplasty: an observational study. Ann R Coll Surg Engl. 2005 Mar;87(2):99-101. doi: 10.1308/147870805X28118. PMID 15826417
- [Background] Elwatidy S, Jamjoom Z, Elgamal E, Zakaria A, Turkistani A, El-Dawlatly A. Efficacy and safety of prophylactic large dose of tranexamic acid in spine surgery: a prospective, randomized, double-blind, placebo-controlled study. Spine (Phila Pa 1976). 2008 Nov 15;33(24):2577-80. doi: 10.1097/BRS.0b013e318188b9c5. PMID 19011538
- [Background] Wong J, Abrishami A, El Beheiry H, Mahomed NN, Roderick Davey J, Gandhi R, Syed KA, Muhammad Ovais Hasan S, De Silva Y, Chung F. Topical application of tranexamic acid reduces postoperative blood loss in total knee arthroplasty: a randomized, controlled trial. J Bone Joint Surg Am. 2010 Nov 3;92(15):2503-13. doi: 10.2106/JBJS.I.01518. PMID 21048170
- [Background] Raveendran R, Wong J. Tranexamic acid reduces blood transfusion in surgical patients while its effects on thromboembolic events and mortality are uncertain. Evid Based Med. 2013 Apr;18(2):65-6. doi: 10.1136/eb-2012-100872. Epub 2012 Aug 4. No abstract available. PMID 22864370
- [Background] Zufferey P, Merquiol F, Laporte S, Decousus H, Mismetti P, Auboyer C, Samama CM, Molliex S. Do antifibrinolytics reduce allogeneic blood transfusion in orthopedic surgery? Anesthesiology. 2006 Nov;105(5):1034-46. doi: 10.1097/00000542-200611000-00026. PMID 17065899
- [Background] Wang H, Shen B, Zeng Y. Comparison of topical versus intravenous tranexamic acid in primary total knee arthroplasty: a meta-analysis of randomized controlled and prospective cohort trials. Knee. 2014 Dec;21(6):987-93. doi: 10.1016/j.knee.2014.09.010. Epub 2014 Oct 23. PMID 25450009
- [Background] Ipema HJ, Tanzi MG. Use of topical tranexamic acid or aminocaproic acid to prevent bleeding after major surgical procedures. Ann Pharmacother. 2012 Jan;46(1):97-107. doi: 10.1345/aph.1Q383. Epub 2011 Dec 27. PMID 22202494

RESULTS

PARTICIPANT FLOW:
Groups:
- Tranexamic Acid: Participants undergoing spinal surgery received a single, topical dose of 3 grams (g) tranexamic acid. The surgeon irrigated the study medication in the wound prior to closure, and aspirated it after five minutes. Drains were placed after the study drug was aspirated.
- Placebo: Participants undergoing spinal surgery received a single, topical dose of matching placebo. The surgeon irrigated the study medication in the wound prior to closure, and aspirated it after five minutes. Drains were placed after the study drug was aspirated.
Period: Overall Study
Arm/Group | Tranexamic Acid | Placebo
Started | 12 | 17
Completed | 12 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Tranexamic Acid: Participants undergoing spinal surgery received a single, topical dose of 3 g tranexamic acid. The surgeon irrigated the study medication in the wound prior to closure, and aspirated it after five minutes. Drains were placed after the study drug was aspirated.
- Total: Total of all reporting groups
Arm/Group | Tranexamic Acid | Placebo | Total
Number analyzed (Participants) | 12 | 17 | 29
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 69 [62 to 72] | 66 [50 to 73] | 68 [60 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 20
  Male | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin Level From Preoperative Appointment to Postoperative Hospital Discharge
Description: Blood loss was calculated from the difference between the level of hemoglobin at the preoperative appointment and the lowest level during the postoperative hospitalization period. Reported here is the change in hemoglobin level after surgery. A negative number indicates a reduction in hemoglobin level.
Time Frame: From preoperative appointment approximately one week before surgery to end of hospital stay up to approximately 5 days after surgery
Population: Only participants, for whom both preoperative and postoperative time points were collected, are reported in this outcome measure.
Measure: Median (Inter-Quartile Range); unit: grams per deciliter (g/dL)
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 11 | 15
grams per deciliter (g/dL) | -3.2 [-4.6 to -2.4] | -4.6 [-5.3 to -4.1]
Statistical Analysis 1: Comparison: Tranexamic Acid vs Placebo; Test type: Superiority; p = 0.1318, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Blood Loss Volume Following Surgery
Description: Blood loss following surgery was defined as the total amount of fluid collected from the drain in the wound site during the hospital stay.
Time Frame: From end of surgery on Day 1 to end of hospital stay up to approximately 5 days
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 12 | 17
mL | 534 [260 to 705] | 530 [320 to 795]

3. Secondary Outcome: Hospital Length of Stay in Days
Description: The number of days the participants stayed in the hospital after surgery was recorded.
Time Frame: From end of surgery on Day 1 to end of hospital stay up to approximately 2 weeks
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 12 | 17
days | 5 [4 to 8] | 6 [5 to 7]

4. Secondary Outcome: Post-operative Blood Transfusions During Hospitalization
Description: All units of blood transfused during the hospital stay after surgery were recorded. One red blood cell unit contains 300 to 360 mL of whole blood.
Time Frame: From end of surgery on Day 1 to end of hospital stay up to approximately 5 days
Measure: Median (Inter-Quartile Range); unit: units of blood
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 12 | 17
units of blood | 0 [0 to 1] | 0 [0 to 1]

ADVERSE EVENTS:
Time Frame: From time of admission to hospital for surgery up to study completion (up to approximately 2.5 years).
Description: Participants were monitored only for the following serious adverse events from time of admission to hospital for surgery up to study completion: myocardial infarction, stroke, thrombosis, and postoperative infection. Non-serious adverse events were not collected in this study.
Arm/Group | Tranexamic Acid | Placebo
Serious Adverse Events (participants affected / at risk) | 3/12 | 1/17
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tranexamic Acid (N=12) | Placebo (N=17)
Myocardial infaction (Cardiac disorders) | 1 (1) | 0 (0)
Postoperative wound infection (Surgical and medical procedures) | 1 (1) | 1 (1)
Postoperative wound infection after release from hospital (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No